CLINICAL TRIAL: NCT05389709
Title: Pharmacy-based Non-interventional Study (NIS) With Iberogast® Advance (STW 5 II).
Brief Title: A Pharmacy-based Observational Study to Learn More About Iberogast Advance in the Real-world Setting
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21970
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Functional Gastrointestinal Disorders Such as Irritable Bowel Syndrome and Functional Dyspepsia; Irritable Bowel Syndrome; Functional Dyspepsia
Keywords: Iberogast Advance
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — iberogast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pharmacy based survey: Patients receive a questionnaire to fill out and return it the Contract Research Organization (CRO) or, alternatively to the pharmacy.
  Interventions: Drug: Iberogast (STW5-II, BAY98-7410)

INTERVENTIONS:
Drug: Iberogast (STW5-II, BAY98-7410) — Survey without any intervention assigned in the study.
  Other Names: Iberogast® Advance

SUMMARY:
This is an observational study in which data from people with functional gastrointestinal disorders who decide on their own or by recommendation of their doctors or pharmacists to take Iberogast Advance are collected and studied. In observational studies, only observations are made without specified advice or interventions.

Functional stomach and bowel (or gastrointestinal) disorders are conditions in which the functionality of the gut, mainly the gut muscles or the gut/brain axis, is disturbed. Functional stomach and bowel disorders cause symptoms like heartburn, cramps and pain of the upper and middle part of the belly, also known as functional dyspepsia (FD) and irritable bowel syndrome (IBS). IBS affects predominantly the lower digestive system and causes symptoms like pain of the belly, cramps, bloating, diarrhea, and constipation.

Iberogast Advance is already available in German pharmacies without prescription for patients with gastrointestinal disorders such as FD and IBS. It contains herb extracts that work against inflammation, are calming, and protect the mucosa (innermost layer of the gastrointestinal tract). Earlier controlled studies with Iberogast Advance have shown how well it works and how it affects the body. Since Iberogast Advance is only available since October 2020, there is no information on its use in the real-world setting yet.

Therefore, the study researchers want to collect data on the use of Iberogast Advance in the real-world setting.

To do this, people with long-term and repeated functional gastrointestinal symptoms who purchase Iberogast Advance from participating pharmacies across Germany will be asked to fill out a questionnaire optionally covering 6 weeks of treatment. The participants will take Iberogast Advance as recommended in the product information.

The main purpose of this study is to see how well Iberogast Advance works and is perceived in the real-world setting. Participants will record how they experience a change of their gastrointestinal symptoms (assessed single-symptom-based) from start and during 6 weeks of treatment. Researchers will then compare the differences and analyze treatment effects.

The researchers will additionally collect information on usage behavior, characteristics of the patients, their symptoms, tolerability and their satisfaction with Iberogast Advance.

There will be no required tests or visits with a study doctor in this study. The researchers will collect the results of the patient questionnaires from Jun 2022 to January 2023.

ELIGIBILITY:
Inclusion Criteria:

* Adult female or male subject aged ≥ 18
* Decision to initiate treatment with Iberogast Advance was made as per pharmacist's routine recommendation practice/by the subject
* Subject purchases Iberogast Advance for his own use
* Not pregnant or lactating
* Not hypersensitive to any of the ingredients of Iberogast Advance

Exclusion Criteria:

* Patients with known hypersensitivity to any of the ingredients of Iberogast Advance
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: German patients who use Iberogast Advance for treatment of gastrointestinal complaints.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Single gastrointestinal symptoms intensity via a five point Likert scale assessed weekly. | Up to 6 weeks
  Patients assessed intensity on 5 point Likert scale as 0=no symptom; 1=mild symptom; 2= moderate symptom; 3=strong symptom; 4= unbearable symptom.

SECONDARY OUTCOMES:
Descriptive analyses of patient characteristics data | At baseline
Descriptive analyses of patient symptoms profile | At baseline
Reason for using Iberogast Advance | At baseline
Long term usage during the previous 6 months | At baseline
Usual dosage applicated assessed weekly | Up to 6 weeks
Onset of noticeable symptom relief after application of Iberogast Advance as assessed by patient weekly. | Up to 6 weeks
Overall treatment effect of Iberogast Advance measured as course of gastrointestinal symptom intensity as assessed by patient | At week 6
Change of symptoms after 6 weeks treatment/observation period via a five point Likert scale | Baseline to week 6
  Patients assessed intensity on 5 point Likert scale as 0=no symptom; 1=mild symptom; 2= moderate symptom; 3=strong symptom; 4= unbearable symptom.
Patients satisfaction as assessed by patients as assessed via a five point Likert scale. | At week 6
  Patients assessed intensity on 5 point Likert scale as 0=no symptom; 1=mild symptom; 2= moderate symptom; 3=strong symptom; 4= unbearable symptom.
Number of participants with gastrointestinal complaints ,categorized by severity. | At week 6
Reason for early termination of Iberogast Advance | At week 6
Tolerability as assessed by the patient | At week 6
  Patients assessed tolerability by using very good; Good; Moderate; Bad; Very bad; Missing values.

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Many Locations, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.